

## Study Title:

A RANDOMIZED OPEN LABEL PHASE II STUDY OF WEEKLY GEMCITABINE PLUS PAZOPANIB VERSUS WEEKLY GEMCITABINE ALONE IN THE TREATMENT OF PATIENTS WITH PERSISTENT OR RELAPSED EPITHELIAL OVARIAN, FALLOPIAN TUBE OR PRIMARY PERITONEAL CARCINOMA

Version Date:

01 February 2017

NCT#:

NCT01610206

 Version: 01Feb2017



# Consent of an Adult to Be in a Research Study

In this form "you" means a person 18 years of age or older who is being asked to volunteer to participate in this study.

| Participant's Name | Medical Record # |
|-----------------------|-------------------------------------------------|
| Principal | Linda R. Duska, M.D. |
| Investigator/Sponsor: | University of Virginia School of Medicine (UVA) |
| | PO Box 800712 |
| | Charlottesville, VA 22908 |
| | Telephone: (434) 982-1719 |
| | Fax: (434) 982-1840 |
| | lduska@virginia.edu |
| Funding Source | Novartis Pharmaceuticals |

# What is the purpose of this form?

This form will provide you with information about this research study. You do not have to be in the study if you do not want to. You should have all your questions answered before you agree to be in this study.

Please read this form carefully. If you want to be in the study, you will need to sign this form. You will be given a signed copy of this form.

# Who is funding this study?

This study is being carried out under the sponsorship of Dr. Linda Duska at the University of Virginia Cancer Center. Some financial support has been provided by Novartis, the manufacturer of pazopanib.

## Why is this research being done?

Chemotherapy is the standard treatment for cancer of the ovary, fallopian tube or peritoneum when it returns after initial treatment. A number of chemotherapy options exist for patients when their cancer grows despite treatment with the most effective chemotherapy (such as carboplatin or cisplatin). One of these chemotherapy agents is gemcitabine.

The purpose of this study is to compare the safety and effectiveness of an experimental drug called pazopanib when given in combination with gemcitabine versus gemcitabine alone for people with ovarian cancer, fallopian tube cancer, or primary peritoneal cancer that has re-grown or not responded after prior treatment.




Gemcitabine in combination with carboplatin is approved for use by the U.S. Food and Drug Administration (FDA) for the treatment of patients with advanced ovarian cancer that has relapsed at least six months after completion of therapy with carboplatin or cisplatin. Gemcitabine is also used as a single agent for cancer of the ovary, fallopian tube or peritoneum when it returns after initial treatment, although this is not an FDA-approved treatment.

Pazopanib is a different kind of chemotherapy drug. Pazopanib works by slowing or stopping the spread of cancer cells by blocking new blood vessel formation. New blood vessel formation is required for tumor growth.

Currently, Pazopanib is approved by the FDA for use in the treatment of patients with advanced kidney cancer and certain types of advanced soft tissue sarcoma (cancer of connective or supportive tissues such as bone, cartilage, fat, muscle...) but has not been approved for use in other cancer types. Pazopanib alone or pazopanib + gemcitabine is NOT approved by the FDA for the treatment of ovarian, fallopian tube, and primary peritoneal cancer. In other words, the combination of pazopanib and gemcitabine is experimental.

You are being asked to take part in this study because you have ovarian cancer, fallopian tube cancer, or primary peritoneal cancer that has regrown or not responded after prior treatment.

Up to 60 people will be in this study at UVA. Approximately 150 people will take part in this study at other institutions in the United States.

# How long will this study take?

You will be required to make weekly office visits while you are receiving study treatment.

You will continue to take pazopanib + gemcitabine or gemcitabine alone as long as there is evidence that your tumor is not growing and you are not experiencing any unacceptable side effects.

After you are finished taking the chemotherapy drug(s), your doctor will ask you to visit the office for follow-up exams every three months for the first two years, every six months for the next year and then yearly for 2 years for a maximum of 5 years.

Your participation in this study will, require an additional 30 minutes during your initial visit with your doctor and an additional 30 minutes during the routine clinical visits you will be making as part of your cancer treatment.




# What will happen if you are in the study?

# SCREENING (will take approximately 1 hour to complete) Visit 1/Day 0

If you agree to participate, you will sign this consent form before any study related procedures take place. Before you can start in the study, there will be a screening period. You will have tests and procedures during this time to make sure you are eligible and it is safe for you to participate. If you have had some of them recently, they may not need to be repeated. This will be up to your study doctor.

# The following exams, tests or procedures are <u>part of regular cancer care</u> and will be done even if you do not join the study:

- History and physical examination which may include pelvic exam. You will also have your heart rate, blood pressure and temperature taken.
- Chest imaging (X-ray or CT scan of the chest)
- A left ventricular ejection fraction (LVEF) test to measure your heart function if you have had prior therapy with a certain type of drug (anthracyclines)
- ECG (tracing of heart waves)-Electrocardiogram to see the electrical activity of your heart.
- CT-scan or MRI of the abdomen and pelvis to measure detectable tumor
- Review of medications and supplements you are currently taking. If you agree to take part in this study, it is very important that you tell your study doctor before starting on this study about all of the medicines you are taking (over-the-counter medications, supplements, prescription medications, or illegal drugs) including any medicines you have taken within the past 2 weeks. The reason this is important is that some medicines can change the way your body handles other medicines and this can increase the risk of side effects. In addition, please talk with the study doctor before you begin taking any new medications or supplements during this study. Your study doctor will look at the medicines you are currently taking to make sure you are allowed to take them on the study. You may be asked to change some of the medicines you are taking. If you need to take a medicine that is not allowed and it cannot be replaced with another medicine, you will not be asked to stop taking it; however, you will not be able to take part in this study.

# The following exams, tests or procedures are not part of regular cancer care and will be <u>done for research</u> purposes:

A urinalysis (testing of urine) to check urine protein levels




- A serum pregnancy test if you are capable of becoming pregnant (this will be done within 14 days prior to receiving study treatment)
- Blood tests to assess blood cell counts; liver and kidney function; blood mineral levels; blood clotting
  function and the CA-125 tumor marker. The amount of blood that will be drawn is approximately 2
  tablespoons. Blood tests to assess thyroid for research purposes will be done on the blood taken as
  part of your routine cancer care. These tests will not require additional blood samples.

If these tests show you are eligible, you will return to the clinic (within 28 days) to begin study treatment.

## **RANDOMIZATION**

Visit 2/Day 1

You will be randomly assigned (like the flip of a coin) to 1 of 2 study treatment groups. You have an equal chance of being assigned to one of the groups. Neither you nor your doctor can choose which study treatment you are assigned. Both you and your doctor will know which of the two groups you are assigned to.

**GROUP 1:** Gemcitabine given as intravenous (IV) infusion (standard of care)

**GROUP 2:** Pazopanib (oral) + Gemcitabine (IV) (Experimental)

Note: Every 21-day period of time is called a cycle.

#### Group 1

Gemcitabine will be put into your vein over 30 minutes, weekly for 2 weeks (Day 1 and Day 8 of each cycle) every 21 days

#### Group2

Gemcitabine will be put into your vein over 30 minutes, weekly for 2 weeks (Day 1 and Day 8 of each cycle) every 21 days

Pazopanib will be taken by mouth daily. Pazopanib should be taken on an empty stomach 1 hour before or 2 hours after meals. The tablets should be swallowed whole and must not be crushed or broken.

**STUDY VISITS** (each visit will last about 60 – 90 minutes):

You will visit your doctor weekly (Day 1 and Day 8 of each cycle) every 21 days. At these visits, you will need the following tests and procedures that are all being done as part of your regular cancer care.




- History and physical examinations which may include a pelvic exam about once every three weeks.
   You will also have your heart rate, blood pressure and temperature monitored at each study visit.
- Blood tests to measure the CA-125 tumor marker blood level prior to each cycle of treatment.
- Chest imaging (X-ray or CT scan of the chest) before the start of every other cycle (i.e. Cycle 2, 4, 6...).as needed
- CT scan or MRI to measure tumor before the start of every other cycle (i.e. Cycle 2, 4, 6...)
- Review of medications you are taking before starting each cycle.
- If you are taking warfarin, your doctor will also check your blood clotting levels.

## The following will be done for research purposes:

 Blood tests to measure blood counts, electrolytes, blood mineral levels, and check liver and kidney function prior to each cycle of treatment (more often if your doctor(s) feels it is needed.)

# In addition, if you are assigned to Group 2, the following tests and procedures will be done for research purposes:

- Blood pressure will be monitored on Day 15 of every cycle; you may do this at home and provide the results to the study doctor or study nurse. (Note blood pressure done on other days will be performed per your regular cancer care).
- An electrocardiogram will be done on Day 1 of cycle 2
- Urine protein levels (UPC) will be examined by urinalysis (testing of urine) before the start of every other cycle (i.e. Cycle 2, 4, 6...).
- You will be given a patient medication calendar to complete throughout the study. The patient medication calendar is a monthly calendar on which you are to record the number of tablet(s) you take each day. You will need to bring the calendar with you to the doctor's office before each cycle, along with any unused study medications and empty medication containers.

#### **FOLLOW UP:**

To monitor your well-being and the status of your cancer, you will undergo these tests and procedures that are part of regular cancer care every 3 months for 2 years and then every 6 months for 1 year and then yearly for 2 years. The maximum follow up period is 5 years:

- History and physical examination which may include pelvic examination CT or MRI scan, if previously detectable tumor was monitored using these methods, as recommended by your physician.
- CA-125 tumor marker blood level as recommended by your physician.
- Chest imaging (X-ray or CT scan of the chest) as recommended by your physician.




## **END OF STUDY:**

After you have completed participation in the study, you will no longer receive the study drug. You, together with your doctor, will determine the next steps in your care plan.

## **Study Schedule:**

Every 21-day period of time is called a cycle. Each cycle is numbered in order. The schedule below shows what will happen to you during Cycle 1 and future cycles as explained previously.

| | | | Cycle 1 | | Cycles | 2+ | | |
|---|---|---|---|---|---|---|---|---|
| | Visit 1 | Day 1 | Day 8 | Day 15 | Day 1 | Day 8 | Day 15 | Follow-up |
| Informed Consent | х | | | | | | | |
| Medical History | Х | | | | х | | | х |
| Physical Exam | Х | | | | х | | | х |
| CT/MRI (if applicable) | Х | | | | х | | | х |
| Chest x-ray (if applicable) | Х | | | | х | | | х |
| ECG | х | | | | x <u>* (</u> Group<br>2 only) | | | |
| Cardiac function (if applicable) | х | | | | | | | |
| Blood draw (for laboratory testing) | x <u>*</u> | x <u>*</u> | x <u>*</u> | | x <u>*</u> | x <u>*</u> | | x<br>(CA-125) |
| Blood pressure | х | х | х | x (Group<br>2 only) | х | х | x (Group<br>2 only) | |
| Heart rate and temperature | х | | х | | х | х | | |
| Urine testing | x <u>*</u> | | | | x <u>*</u><br>(Group 2<br>only, even<br>cycles) | | | |
| Pregnancy test (if applicable) | х | | | | | | | |
| Review side effects | | Х | Х | Х | х | Х | | х |
| Gemcitabine | | Х | Х | | х | Х | | |
| *Pazopanib (Group 2 only) | | Daily | | | | | | |
| *Pill calendar (Group 2 only) | | Х | X | x | х | х | х | |

An \* indicates procedures done for research purposes. All other procedures are performed as part of your clinical care.




## What are your responsibilities in the study?

You have certain responsibilities to help ensure your safety. These responsibilities are listed below:

- You must come to each study visit or notify the study doctor or study staff if you are unable to do so.
- You must be completely truthful about your health history.
- Follow all instructions given.
- You should tell the study doctor or study staff about any changes in your health or the way you feel.
- Ensure that the study drug is taken as instructed, keep the study drug in a safe place away from other children, return any unused study drug at each visit, and report any lost or missed tablets.
- Ensure that the study drug is taken only by you, the person for whom it has been prescribed.
- Answer all of the study-related questions completely.
- You must not eat grapefruit or drink grapefruit juice during the course of your participation in this study.
- Inform the study doctor or study staff as soon as possible if you have to take any new medications, including anything prescribed by a doctor or those that you can buy without a prescription (over-thecounter), including herbal supplements and vitamins. The study doctor will let you know if you can take these medications.

## If you want to know about the results before the study is done:

During the study your study leader will let you know of any test results that may be important to your health. In addition, as the research moves forward, your study leader will keep you informed of any new findings that may be important for your health or may help you decide if you want to continue in the study. The final results of the research will not be known until all the information from everyone is combined and reviewed. At that time you can ask for more information about the study results.

# What are the risks of being in this study?

Research studies often involve some risks. You should talk to your study doctor about any side effects that you have while taking part in the study. The risks of this study are as follows:

### Risks and side effects related to the **Gemcitabine** include those which are:

## Likely:

 Low white blood cell counts that could lead to infection

- Low red blood cell counts that could cause anemia
- Mild nausea




- Fatigue
- Hair loss

#### **Less Likely**

- Flu-like symptoms such as fatigue, muscle aches, fever lasting 1-2 days after gemcitabine treatments
- Infection requiring treatment with medicines
- Low platelets that could lead to bleeding
- Nausea and vomiting
- Diarrhea or constipation
- Mouth sores may occur; you will be given treatment to make them more tolerable.
   Mouth sores improve over time.

- Numbness or tingling in the hands and/or feet
- Abnormalities in the blood tests that measure liver function
- Fluid retention in the feet, legs, and weight gain
- Kidney function abnormalities, with the appearance of protein or blood in the urine
- Rash may occur, involving the body and/or legs.
- Changes in taste, or a metallic taste

#### Rare but serious

- Confusion, hearing problems, heart failure, abnormal heart rhythms, high blood pressure, low blood
  pressure, blood clots in the legs or lungs, bowel obstruction, bleeding, severe infections leading to
  death. The relationship of these events to the administration of the chemotherapy drugs has not been
  proven, since all patients who have received these drugs have underlying cancer, which may cause
  some or all of these effects by itself.
- Rarely, severe lung damage has occurred in patients being treated with the combination of gemcitabine and docetaxel. In most cases the lungs got better when the treatments were stopped.
- Rarely, a condition affecting the blood and kidneys called hemolytic uremic syndrome has occurred. When this happens the kidney damage can sometimes be permanent.

#### Risks and side effects related to **Pazopanib**:

As of 9 September 2016, about 5919 patients and healthy volunteers had received pazopanib (either as monotherapy or in combination) out of more than <u>8746</u> patients enrolled in oncology, ophthalmology, and psoriasis studies. Pazopanib can cause side effects, although not everybody gets them. Some side effects can be life-threatening or fatal. The side effects below are those reported by patients who have taken pazopanib either in a clinical trial or as prescribed by their doctors. The side effects are listed according to the highest number of patients who had them in pazopanib studies, as very common, common, or uncommon. Not all side effects of pazopanib are known and further studies are under way. If you experience one or more side effects, please speak with your study doctor.




## Very common side effects occurring in greater than 10 out of 100 subjects included:

- Increase in blood sugar
- Stomach pain or discomfort
- Diarrhea
- feeling or being sick ( nausea, vomiting, abdominal pain/discomfort)
- loss of strength and energy, weakness
- loss of appetite
- changes in hair color
- high blood pressure
- headache
- weight loss
- unusual hair loss or thinning
- A skin reaction or pain on the palms of the hands or soles of the feet (including tingling, numbness, pain, swelling or reddening.
- Loss of skin pigment
- chest pain
- problems with taste
- mouth sores/inflammation of the lining in the mouth

- cough
- shortness of breath
- dizziness
- exfoliative rash (rash with skin peeling)
- muscle pain
- pain in the bones, muscles, ligaments, joints and tendons
- swelling caused by fluid in the, hands, ankles, or feet
- slow heart rate
- increase in some substances (enzymes)
   produced by the liver. This may show up
   in your blood tests. Patients over 60
   years of age may be at greater risk of an
   increase of one of the enzymes, called
   ALT.
- decrease in albumin (a protein found in the blood; may indicate a disruption of liver function)

## Common side effects occurring in between 1 and 10 out of 100 subjects included:

- hoarse voice
- blurry vision
- heartburn (indigestion)
- nosebleeds
- blood in the urine
- low white blood cell counts (the cells which fight infection)
- a decrease in the number of cells involved in blood clotting
- protein in the urine (a sign that kidneys are not working normally)

- under active thyroid gland (a gland important in regulating metabolism)
- abnormal liver function
- increase in lipase (an enzyme from the pancreas); may be a sign of a pancreas problem
- changes in heart's electrical conduction (QT-prolongation)
- temporary reduction in blood supply to the brain (mini-stroke)
- reduction of blood supply to the heart (angina)




- sudden collapse of the lung
- heart becomes less effective at pumping blood (cardiac dysfunction)
- chest pain, shortness of breath, leg pain, and swelling of the legs/feet. These could be signs of a blood clot in your body (thromboembolism). If the clot breaks off, it may travel to your lungs and this may be life threatening or even fatal
- severe bleeding in the lungs
- heart attack
- chills
- skin rash
- dry skin
- nail disorder

- excessive stomach or intestinal gas (flatulence)
- muscle spasms
- increase in bilirubin (substance produced by the liver; may indicate a disruption of liver function)
- increase in gamma-glutamyl transpeptidase (a liver enzyme; may indicate a disruption of liver function)
- •
- severe bleeding in digestive tract (stomach and intestine) and brain
- infection, with or without changes in white blood cells (cells that fight infection)

#### Uncommon side effects occurring in less than 1 out of 100 subjects included:

- Severe bleeding in the brain
- a dangerous rapid fluttering of the heart (Torsades de Points)
- hole in the gut wall (perforation)
- abnormal connection between parts of the digestive tract (fistula)
- stroke
- liver failure (which could possibly result in death)
- a sudden and severe rise in blood pressure (hypertensive crisis)
- inflammation of the pancreas

- Separation or tear of the lining of the back part of the eye (retinal detachment or tear). This can result in blurry or impaired vision.
- Abnormal increase in the number of red blood cells (polycythemia)
- Blood clots accompanied by a decrease in red blood cells and cells involved in clotting. These clots may harm organs such as the brain and kidneys.

#### Rare Side Effects (These may affect up to 1 in 1000 people):

- Swelling of the brain that may be associated with high blood pressure, headache, loss of speech or vision, and/or seizure, which may be life threatening
- Scarring of the lung tissue, leading to lung stiffness, affecting the ability to breathe (Interstitial Lung Disease) and inflammation of the lung tissue (pneumonitis), which can be fatal.




### Other Risks of Pazopanib

One patient developed liver failure and died shortly after beginning treatment with the combination of gemcitabine and pazopanib.

Lung infection has been observed in 1 out of 1000 patients treated with pazopanib.

Neutropenia (low white blood cell count), thrombocytopenia (decrease in the number of cells involved in blood clotting), and palmar-plantar erythrodysaethesia syndrome (hand-foot syndrome) were observed more frequently in patients of East Asian descent.

Patients who carry a specific gene (HLA B\*57:01 allele) have an increased chance of abnormal liver function (ALT elevations) due to Pazopanib.

Studies in animals indicate that pazopanib may slow or stop bone growth. There is a possibility that pazopanib may affect bone growth in children, adolescents and young adults who are still growing.

Severe and fatal liver disease has occurred in patients treated with pazopanib and patients older than 65 years are at greater risk for this. During this study, blood tests will be checked to look for liver injury. People with liver injury may feel very tired, or sick and not want to eat, have yellow skin or eyes, and they may also develop rash or fever.

During this study, blood tests will be checked to look for liver injury. People with liver injury may feel very tired or sick and not want to eat, have yellow skin or eyes, and they may also develop rash or fever.

Let your doctor know if you have any of these symptoms, especially if your doctor says you have abnormal liver blood tests. If your doctor finds that your blood tests suggest liver injury that is not severe, your doctor may recommend you continue taking pazopanib and may ask you to stop taking other drugs which may cause liver injury. Blood tests (about 1/3 tablespoon of blood per test) for possible liver injury will be repeated every week until they get better. These tests will be done per your clinical care.

If your blood tests get worse, your doctor may tell you to stop taking pazopanib altogether. If you have a liver injury from pazopanib, it will usually heal when pazopanib is stopped. It is possible that a small number of people may continue to have liver injury after they stop taking pazopanib.

If you are to have surgery, please speak with your doctor because pazopanib may affect wound healing.




There may be other side effects that may happen that are not known now. For example, all drugs can cause an allergic reaction in some patients. Certain problems can become worse if not treated quickly. Call the study doctor right away if: <Amend list below, as required>

- You feel very tired or faint
- You feel pain or sick in your stomach and you do not want to eat
- You bruise easily or develop itching
- You have yellow eyes or skin, or dark urine
- You become confused.

If you experience certain other serious problems (such as an allergic reaction, swelling, difficulty breathing, a bad skin rash, liver or kidney damage, or changes in your heart rhythm), you may be asked to return to the clinic for more tests. This may include more blood tests. The study doctor will explain these tests to you if they are needed. You may also need to stop taking the study drug after talking with the study doctor.

### **Risks of Sharing the Drug**

Do not share the study drug with anyone. It is prescribed only for you and could hurt someone else. Keep it out of reach of children and people not able to read or understand the label.

#### **Blood Donation**

If you participate in this study it may affect your ability to donate blood. If you have any questions call the organization where you donate blood and talk to one of their nurses.

## Risks of having your blood drawn:

Having blood drawn may cause:

- pain (common),
- a bruise (sometimes),
- fainting or passing out (not very often), and
- infection (rare).

If the people doing the study are exposed to your blood or body fluids in a way that could give them a disease, your blood may be tested. The tests might check for:

- hepatitis,
- HIV (Human Immunodeficiency Virus), or
- other infections.




You and the person exposed would be told the test results. However, your name would be kept private. If your test is positive for hepatitis or HIV or any other infection that may affect your clinical care, we will tell you the results and help you understand what the results mean for you.

## **Risks for women: Pregnancy and Contraception**

The drug(s) used in this study can harm an unborn or nursing baby. Therefore, you cannot be in this study if you are pregnant or nursing a baby. A pregnancy blood test will be done about 14 days before receiving any study treatment if you are a woman able to become pregnant as part of your clinical care. This test must be negative in order to continue study participation.

It is important you understand that if you could become pregnant, you need to use birth control while on this study. You and your partner must use an approved form of birth control during this study. Examples of birth control you may use are:

- Norplant
- IUD (intrauterine device)
- Depo-Provera

- Birth Control Pills
- Birth Control Patch
- Sterilization

The birth control methods listed below are less effective. They may be used if combined with other birth control methods:

- Condoms
- Jellies or foam
- Withdrawal
- Sponge

- Diaphragm
- Rhythm
- Cervical cap

Ask your doctor for more details about the proper birth control method for you. If you become pregnant during this study, you must tell your doctor right away. Your doctor will discuss your treatment and the effect on the pregnancy.

As outlined earlier, there are certain medications and supplements that may interact with the study drug(s). You should not take any new medications or supplements without discussing it with your study doctor first.

For more information about risks and side effects, ask your study doctor.

#### Other unexpected risks:

You may have side effects that we do not expect or know to watch for now. Call the study leader if you have any symptoms or problems.




# Could you be helped by being in this study?

We cannot promise that you will be helped by being in this study.

You may or may not benefit from being in this study. Possible benefits include: treatment with pazopanib + gemcitabine may be more effective in treating your cancer compared to gemcitabine alone, however, there is no proof of this yet. In addition, information researchers get from this study may help others in the future.

# What are your other choices if you do not join this study?

You do not have to be in this study to be treated for your illness or condition. You can receive the usual treatment even if you choose not to be in this study. If you do not take part in this study, your other choices may include:

- Getting standard treatment or care for your cancer without being in a study. Other treatments include chemotherapy such as gemcitabine, other forms of immunotherapy, radiotherapy, or surgery, alone or in combination
- Taking part in another study
- Getting no treatment
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

Talk to your doctor about your choices before you decide if you will take part in this study.

If you are an employee of UVa your job will not be affected if you decide not to participate in this study. If you are a student at UVa, your grades will not be affected if you decide not to participate in this study.

## Will you be paid for being in this study?

You will not get any money for being in this study.

# Will being in this study cost you any money?

The following procedures/tests, which are being done only for research purposes, will be provided at no cost to you or your health insurance: The cost of the drug pazopanib, urinalysis, thyroid, liver function tests, ECG on Day 1 of Cycle 2, and blood pressure test on Day 15 of each cycle.

You and/or your insurance company must pay for any tests or care given beyond what is required in this study. In addition, you and/or your health insurance may also have to pay for other drugs or treatments that are given to help you control any side effects. You will have to pay for any costs not covered by your health plan. You may be responsible for any co-payments or deductibles. You may wish to ask for an estimate of your 




financial costs. You may also wish to check with your insurance company before the study starts. Ask what they will cover and if they require you to get their permission before you decide to be in the study.

You will be responsible for the cost of travel to come to any study visit and for any parking costs.

## What if you are hurt in this study?

You do not give up any legal rights, such as seeking compensation for injury, by signing this form. If you feel you have been injured as a result of this study you may contact the Principal Investigator or the IRB (phone numbers are located near the end of this form). If you are hurt as a result of being in this study, there are no plans to pay you for medical expenses, lost wages, disability, or discomfort. The charges for any medical treatment you receive will be billed to your insurance. You will be responsible for any amount your insurance does not cover.

# What happens if you leave the study early?

You can change your mind about being in the study any time. You can agree to be in the study now and change your mind later. If you decide to stop, please tell us right away. You do not have to be in this study to get services you can normally get at the University of Virginia.

Even if you do not change your mind, the study leader can take you out of the study. Some of the reasons for doing so may include

- a) Your study physician is concerned about your health
- b) Your condition gets worse
- c) The side effects of the treatment are too dangerous for you
- d) New information shows the study treatment will not work or is not safe for you
- e) You do not follow your doctor's instructions
- f) The study sponsor closes the study for safety, administrative or other reasons

## How will your personal information be shared?

The UVa researchers are asking for your permission to gather, use and share information about you for this study. If you decide not to give your permission, you cannot be in this study, but you can continue to receive regular medical care at UVA.

## If you sign this form, we may collect any or all of the following information about you:

o Personal information such as name, address and date of birth




 Your health information if required for this study. This may include a review of your medical records and test results from before, during and after the study from any of your doctors or health care providers. This may include mental health care records, substance abuse records, and/or HIV/AIDS records.

## Who will see your private information?

- The researchers to make sure they can conduct the study the right way, observe the effects of the study and understand its results
- o People or groups that oversee the study to make sure it is done correctly
- o The sponsor(s) of this study, and the people or groups it hires to help perform or review this research
- Insurance companies or other organizations that may need the information in order to pay your medical bills or other costs of your participation in the study
- Tax reporting offices (if you are paid for being in the study)
- People who evaluate study results, which can include sponsors and other companies that make the drug or device being studied, researchers at other sites conducting the same study, and government agencies that provide oversight such as the Food and Drug Administration (FDA) if the study is regulated by the FDA.
- o If you tell us that someone is hurting you, or that you might hurt yourself or someone else, the law may require us to let people in authority know so they can protect you and others.

Some of the people outside of UVa who will see your information may not have to follow the same privacy laws that we follow. They may release your information to others, and it may no longer be protected by those laws.

The information collected from you might be published in a medical journal. This would be done in a way that protects your privacy. No one will be able to find out from the article that you were in the study.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

What if you sign the form but then decide you don't want your private information shared? You can change your mind at any time. Your permission does not end unless you cancel it. To cancel it, please send a letter to the researchers listed on this form. Then you will no longer be in the study. The researchers will still use information about you that was collected before you ended your participation.

A copy of this consent form will be put in your medical record. (This is not the same as the record of this research study.) This means that everyone who is allowed to see your medical records will be able to find out that you are in this study. This is done so your regular doctors will know what you receive as part of this study. If you have other health problems during the study, they will be able to treat you properly.




## Please contact the researchers listed below to:

- Obtain more information about the study
- Ask a question about the study procedures or treatments
- Report an illness, injury, or other problem (you may also need to tell your regular doctors)
- Leave the study before it is finished
- Express a concern about the study

### **Principle Investigator**

Linda R. Duska, M.D. University of Virginia School of Medicine (UVA) PO Box 800712 Charlottesville, VA 22908

Telephone: (434) 982-1719 Iduska@virginia.edu

## What if you have a concern about this study?

You may also report a concern about this study or ask questions about your rights as a research subject by contacting the Institutional Review Board listed below.

University of Virginia Institutional Review Board for Health Sciences Research PO Box 800483

Charlottesville, Virginia 22908 Telephone: 434-924-9634

When you call or write about a concern, please give as much information as you can. Include the name of the study leader, the IRB-HSR Number (at the top of this form), and details about the problem. This will help officials look into your concern. When reporting a concern, you do not have to give your name.

# **Signatures**

### What does your signature mean?

Before you sign this form, please ask questions about any part of this study that is not clear to you. Your signature below means that you have received this information and all your questions have been answered. If you sign the form it means that you agree to join the study. You will receive a copy of this signed document.


| PARTICIPANT | PARTICIPANT | <br>DATE | |
|---|---|---|---|
| (SIGNATURE) | (PRINT) | DATE | |
| To be completed by participant i | f 18 years of age or older. | | |
| • | above – leave this line blank. Instea | bject does not speak English well or at all, th<br>ad, the participant should sign the Short Forn | |
| Daniel Oktobalia Communi | | | |
| | | study to the potential subject, allowed have answered all their questions. | them |
| By signing below you confirm tha | | • | them |
| By signing below you confirm that time to read the consent or have PERSON OBTAINING CONSENT | PERSON OBTAINING CONSENT | have answered all their questions. | them |

## **Consent from Impartial Witness**

If this consent form is read to the subject because the subject is blind or illiterate, an impartial witness not affiliated with the research or study doctor must be present for the consenting process and sign the following statement. The subject may place an X on the Participant Signature line above.

If an interpreter was used to explain this study to a potential subject, the interpreter must sign and date the

DATE

INTERPRETER

(PRINT)


**INTERPRETER** 

(SIGNATURE)

line above.



I agree the information in this informed consent form was presented orally in my presence to the **identified individual(s)** who has had the opportunity to ask any questions he/she had about the study. I also agree that the **identified individual(s)** freely gave their informed consent to participate in this trial.

| Subject | the identified individual(s): | |
|-------------------------------|-------------------------------|------|
| IMPARTIAL WITNESS (SIGNATURE) | IMPARTIAL WITNESS (PRINT) | DATE |
